CLINICAL TRIAL: NCT01993472
Title: Andrographolides With or Without Capecitabine for Elderly Patients With Locally Advanced or Recurrent or Metastasis Inoperable Colorectal Cancer: a Randomized, Open-label Trial.
Brief Title: Study of Andrographolides With or Without Capecitabine to Treat Colorectal Cancer
Acronym: AGCRC-013
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual rate
Sponsor: Gu Yanhong (Other)
Responsible Party: Sponsor-Investigator, Gu Yanhong, Director, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGCRC-013; ANDRO-JSPPH-2013 (Other: Jiangsu Province People's Hospital)
Record Dates: First submitted 2013-11-12; First posted 2013-11-25 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Andrographolides with Capecitabine (Experimental): Capecitabine1250mg/m2 , bid，d1-14，q3w, Andrographolides 500mg，qd，d1-14，q3w;
  Interventions: Drug: Andrographolides; Drug: Capecitabine
- Capecitabin alone (Active Comparator): Capecitabine1250mg/m2 , bid，d1-14，q3w,
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Andrographolides — comparison of efficacy of Andrographolides combined with Capecitabine or Capecitabine alone in treatment of colorectal cancer
  Other Names: xiyanpingzhusheye
  Arms: Andrographolides with Capecitabine
Drug: Capecitabine
  Other Names: Xeloda

SUMMARY:
The purpose of this study is to determine the efficacy and safety of Andrographolides combined with Capecitabine in treatment of elderly patients with locally advanced or recurrent or metastasis inoperable colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of adenocarcinoma of the colon or rectum
2. Locally advanced or recurrent or metastasis inoperable disease
3. At least 1 measurable or non-measurable lesion per RECIST version 1.1 guidelines. Lesion must not be chosen from a previously irradiated field unless there had been documented tumor progression in that lesion prior to randomization. All sites of disease must be evaluated ≤ 28 days prior to randomization.
4. Man or woman ≥ 65 years of age
5. Hematological function, as follow: (≤ 10 days prior to randomization)

   * Absolute neutrophil count (ANC) ≥ 1.5×109/L
   * Platelet count ≥ 75×109/L
   * Hemoglobin ≥ 8.0 g/dL
6. Renal function, as follows: (≤ 10 days prior to randomization)

   * Creatinine≤ 1.5×ULN
7. Hepatic function, as follow: (≤ 10 days prior to randomization)

   * Aspartate aminotransferase (AST) ≤ 3×ULN(if liver metastases≤ 5×ULN )
   * Alanine aminotransferase (ALT) ≤ 3×ULN(if liver metastases≤ 5×ULN )
   * Total bilirubin≤ 1.5×ULN
8. Subject or subject's legally acceptable representative has provided informed consent

Exclusion Criteria:

1. Symptomatic brain metastases requiring treatment
2. History of other malignancy, except:

   * Malignancy treated with curative intent and with no known active disease present for ≥ 5 years prior to randomization and felt to be at low risk for recurrence by the treating physician
   * Adequately treated non-melanomatous skin cancer or lentigo maligna without evidence of disease
   * Adequately treated cervical carcinoma in situ without evidence of disease
   * Prostatic intraepithelial neoplasia without evidence of prostate cancer
3. Antitumor therapy(eg, chemotherapy, hormonal therapy, immunotherapy, antibody therapy) ≤ 21 days before randomization. Subjects must have recovered from any acute radiotherapy-related toxicity
4. Radiotherapy≤ 14 days before randomization. Subjects must have recovered from any acute radiotherapy-related toxicities
5. Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia)≤ 6 months prior to randomization
6. History of interstitial lung disease(ILD) eg, interstitial pneumonitis, pulmonary fibrosis or evidence of ILD on baseline chest CT or MRI
7. History of any medical or psychiatric condition or labortory abnomality that in the opinion of the investigator may increase the risk associated with the study participation or investigational product administration or may interfere with the interpretation of the results
8. Unstable pulmonary embolism, deep vein thrombosis, or other significant arterial/venous thromboembolic event ≤ 30 days before randomization. If on anticoagulation, subject must be on stable therapeutic dose prior to rangdomization.
9. Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures or is unwilling or unable to comply with study requirements

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From date of randomization until the date of first documented progression，assessed up to 100 months

SECONDARY OUTCOMES:
overall survival | From date of randomization until the date of death from any cause，assessed up to 100 months
Response Rate | From date of randomization until the date of first documented partial response or complete response, assessed up to 100 months
Quality of Life | From date of randomization until the date of death from any cause，assessed up to 100 months

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Bruchard M, Mignot G, Derangere V, Chalmin F, Chevriaux A, Vegran F, Boireau W, Simon B, Ryffel B, Connat JL, Kanellopoulos J, Martin F, Rebe C, Apetoh L, Ghiringhelli F. Chemotherapy-triggered cathepsin B release in myeloid-derived suppressor cells activates the Nlrp3 inflammasome and promotes tumor growth. Nat Med. 2013 Jan;19(1):57-64. doi: 10.1038/nm.2999. Epub 2012 Dec 2. PMID 23202296